CLINICAL TRIAL: NCT07106229
Title: A Phase 3, Multicentre, Randomised, Double Blind, Placebo-controlled Study to Evaluate the Effectiveness, Safety, and Tolerability of MAG200 (an Allogeneic Adipose-derived Mesenchymal Stem Cell Preparation) Administered by Intra-articular Injection to Adult Participants With Symptomatic Osteoarthritis of the Knee.
Brief Title: A Study to Investigate the Effectiveness, Safety, and Tolerability of MAG200 Solution for Intra-articular Injection Compared With Placebo in Participants Aged 35 to 75 Years of Age With Symptomatic Osteoarthritis of the Knee.
Acronym: nexcell-OAK
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Magellan Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-OAK-003
Record Dates: First submitted 2025-07-15; First posted 2025-08-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthristis
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomised to receive placebo, or MAG200 at a dose of 20 million cells (20M), or MAG200 at a dose of 100 million cells (100M).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- 20M MAG200 (Experimental): Participants in this arm will receive MAG200 at a dose of 20 million cells (20M).
  Interventions: Biological: allogeneic human adipose-derived mesenchymal stem cells
- 100M MAG 200 (Experimental): Participants in this arm will receive MAG200 at a dose of 100 million cells (100M)
  Interventions: Biological: allogeneic human adipose-derived mesenchymal stem cells

INTERVENTIONS:
Biological: allogeneic human adipose-derived mesenchymal stem cells — The Investigational Product MAG200 is a preparation of 5 mL allogeneic human adipose-derived mesenchymal stem cells (MSCs).
  Arms: 100M MAG 200; 20M MAG200
Other: Placebo — Placebo is commercially available injectable normal saline (0.9% Sodium Chloride in Water for Injection)
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm whether MAG200 (20M or 100M) will improve pain and function of participants with osteoarthritis of the knee compared with placebo. In addition, the two strengths of MAG200 will be compared.

In this study, participants will receive a single injection of placebo or allogeneic ADMSCs (MAG200) administered by IA injection. Participants will be randomised to receive placebo, or MAG200 at a dose of 20 million cells (20M), or MAG200 at a dose of 100 million cells (100M).

It is anticipated that the study will run for approximately 48 months.

ELIGIBILITY:
Inclusion Criteria

1. Males and females aged ≥ 35 years to ≤ 75 years inclusive.
2. BMI ≥ 19.0 to ≤ 35.0 kg/m2.
3. Documented clinical diagnosis of OA of the study knee.
4. Documented radiological grading of Grade 2 or Grade 3 medial and/or lateral compartment OA of the study knee.
5. Documented radiological grading of OARSI JSN 1-2 of the medial and/or lateral compartment of the study knee.
6. Primary OA treatment of the study knee already attempted within the last 12 months, defined as:

   1. Prescribed analgesia/anti-inflammatory medication where appropriate, AND
   2. an attempted exercise program prescribed by a physical therapist (e.g., physiotherapist, osteopath) or medical practitioner for at least 8 weeks, AND
   3. weight management, where appropriate.
7. Moderate to severe knee specific activity related pain score on the NRS for Pain over the past week.
8. Moderate to severe knee specific functional limitation on KOOS-PS.
9. Less than 5 degrees varus or valgus knee deformity of the study knee relative to neutral alignment.

Exclusion Criteria

1. Any of the following relating to the study knee:

   1. Radiological evidence of KL Grade 4 OA (involving medial, lateral and/or patellofemoral compartment) or OARSI JSN 3.
   2. History of recurrent mechanical instability and / or locking.
   3. Joint surgery or significant knee injury within 12 months prior to Day 1.
   4. Metal in-situ resulting in metal artefact which impacts/prevents MRI assessment.
   5. MRI confirmed:

   i. Generalised full thickness chondral loss involving tibial and/or femoral weight bearing surfaces ii. Total meniscectomy iii. Complete posterior meniscal root tear iv. Subchondral insufficiency fracture v. Osteonecrosis vi. Malignant bone marrow infiltration vii. Solid tumors viii. Traumatic fracture/bone contusion ix. Knee pathology requiring orthopaedic assessment/intervention (e.g., significant loose body)
2. Other causes of the knee symptoms unrelated to knee OA.
3. Significant and debilitating OA in the non-study knee.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of MAG200 on osteoarthritis pain and function | 12 months
  Co-primary endpoints:
  * Change from baseline in pain by Knee Injury and Osteoarthritis Outcome Score pain subscale (KOOS Pain): 0-100 scale (0=extreme knee pain, 100=no knee pain)
  * Change from baseline in function as measured by Knee Injury and Osteoarthritis Outcome Score function in daily living subscale (KOOS-ADL): 0 to 100 scale (0=extreme knee problems, 100=no knee problems)

SECONDARY OUTCOMES:
To assess the effect of MAG200 on osteoarthritis pain | 1, 3, 6, 9, and 12 months
  Change from baseline in activity related pain assessed using an 11-point (0 to 10) Numeric Rating Scale (NRS) (0=no pain, 10=extreme pain)
To assess the response rate of MAG200 | 1, 3, 6, 9, and 12 months
  Response according to OMERACT-OARSI (Outcome Measures in Rheumatology - Osteoarthritis Research Society International) Responder Analysis.
  OMERACT-OARSI response is defined as either 1) improvement in pain or physical function ≥ 50% and an absolute change ≥ 20 points on a 0-100 scale; or 2) improvement of ≥ 20% and with an absolute change ≥ 10 points on a 0 to 100 scale in at least two of the following three categories: pain, physical function, and patient's global assessment of osteoarthritis activity.
To assess the effect of MAG200 on radiological progression | 12 months
  Change from baseline in articular cartilage thickness assessed by quantitative MRI

OTHER OUTCOMES:
Adverse event reporting | Baseline to 12 months
  Incidence of treatment emergent adverse events

IPD SHARING:
Plan to Share IPD: Yes
Outcome data of published/reported results
Time Frame: Individual de-identified participant data which underlie results reported in this article will be available upon publication. Material will be accessible to investigators whose proposed use of data has been approved by an independent review committee and for data meta-analysis. Requests are to be directed to the corresponding author of the article. No end date is given for request of data.
Access Criteria: Requests are to be directed to the corresponding author of the article (clinicaltrials@magellanstemcells.com.au)